CLINICAL TRIAL: NCT04616560
Title: A Phase 2 Study of DS-8201a (NSC# 807708) in Adolescents, or Young Adults With Recurrent HER2+ Osteosarcoma
Brief Title: Trastuzumab Deruxtecan for the Treatment of HER2+ Newly Diagnosed or Recurrent Osteosarcoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - Stage 1 has met accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-08428; NCI-2020-08428 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UM1CA228823 (NIH); PEPN1924 (Other: Pediatric Early Phase Clinical Trial Network); PEPN1924 (Other: CTEP)
Record Dates: First submitted 2020-11-04; First posted 2020-11-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Osteosarcoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Specimen Handling; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (trastuzumab deruxtecan) (Experimental): Patients receive trastuzumab deruxtecan IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 35 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography or MUGA, blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516

SUMMARY:
This phase II trial studies the effects of trastuzumab deruxtecan in treating patients with HER2 positive osteosarcoma that is newly diagnosed or has come back (recurrent). Trastuzumab deruxtecan is in a class of medications called antibody-drug conjugates. It is composed of a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug, called deruxtecan. Trastuzumab attaches to HER2 positive tumor cells in a targeted way and delivers deruxtecan to kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the proportion of patients with recurrent measurable osteosarcoma treated with trastuzumab deruxtecan (DS-8201a) who are event free (%EF) at 24 weeks.

SECONDARY OBJECTIVES:

I. To assess the safety of DS-8201a in patients with recurrent osteosarcoma. II. To describe the pharmacokinetics of DS-8201a in patients with recurrent osteosarcoma.

III. To estimate the objective response rate (ORR), event free survival (EFS), overall survival (OS) and duration of response (DOR) of patients with recurrent, measurable osteosarcoma.

EXPLORATORY OBJECTIVES:

I. To describe the relationship between potential biomarkers and response to DS-8201a.

II. To evaluate quantitative circulating tumor deoxyribonucleic acid (DNA) (ctDNA) and circulating tumor cells (CTCs) as a surrogate markers of response in recurrent osteosarcoma.

OUTLINE:

Patients receive trastuzumab deruxtecan intravenously (IV) over 30-90 minutes on day 1. Treatment repeats every 21 days for 35 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography or multigated acquisition scan (MUGA), blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 12 years and =< 39 years of age at the time of study enrollment
* Patients must have had histologic verification of osteosarcoma at original diagnosis or relapse

  * Patients with diagnoses of osteosarcoma and confirmed HER2 expression of > 10% of osteosarcoma cells are eligible for the intervention

    * Note: There is a mandatory tissue submission for HER2 staining during the Step 0 Eligibility Screening process. Metastatic tissue, when possible from the most recent relapse, is strongly preferred for HER2 staining over archival tissue from primary resection or diagnostic biopsy. The evaluation period for HER2 staining to determine eligibility for therapy will be less than 4 weeks from screening enrollment
* Patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Patients with clinically inactive brain metastases may be included in the study. Patients with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. Lastly, patient must have unresectable lesions or lesions with no intention to surgically remove in the 6 months following enrollment
* Patient's current disease state must be one for which they have received at least standard initial therapy, defined as systemic therapy combined with either radiation or surgery for local control of the primary tumor at diagnosis. Prior therapy after relapse is not required
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0 or 1. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age. Patients who are non-ambulatory as a result of prior surgical treatment for osteosarcoma should be considered ambulatory for the purposes of assessing performance status
* Patients must have recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met, e.g., blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive: For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment

    * >= 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent
  * Antibodies: >= 4 weeks (28 days) must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * Corticosteroids
  * Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Stem cell Infusions (with or without total body irradiation [TBI]):

    * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion and no evidence of graft versus host disease (GVHD)
    * Autologous stem cell infusion including boost infusion: >= 30 days
  * Vellular therapy: >= 30 days after the completion of any type of cellular therapy (e.g., modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Radiation therapy (XRT)/external beam irradiation including protons: >= 4 weeks (28 days) including palliative radiation therapy to the chest. >= 14 days after palliative local XRT to areas other than the chest or for whole brain radiotherapy
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, samarium): >= 42 days after systemically administered radiopharmaceutical therapy
  * Patients must not have received prior HER2 therapies including antibody drug conjugates (e.g. TDM-1 or DS-8201a), HER2 directed cellular therapies, HER2 receptor therapy (e.g. trastuzumab, pertuzumab) or small molecule antagonists of HER2 (e.g lapatinib or neratinib)
* Patients must be at least 7 days from the date of last surgery
* Peripheral absolute neutrophil count (ANC) >= 1000/mm^3, (granulocyte colony-stimulating factor [G-CSF] administration is not allowed within 1 week prior to Step 1 screening assessment) (for patients with solid tumors without known bone marrow involvement)
* Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment) (for patients with solid tumors without known bone marrow involvement)
* Hemoglobin >= 8.0 g/dL at baseline (Red Blood Cell transfusion is not allowed within 1 week prior to screening assessment) (for patients with solid tumors without known bone marrow involvement)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age: 12 to < 13 years; Maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
  * Age: 13 to < 16 years; Maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: >= 16 years; Maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)

    * For participants less than 18 years of age that screen fail only based on creatinine, a 24 hour urine collection may be used instead to confirm eligibility. A calculated GFR > 60 mL/min/1.73 m^2 using a 24 hour collection will meet criteria for inclusion on this trial
* Bilirubin (sum of conjugated + unconjugated or total) =< 1.5 x upper limit of normal (ULN) for age. For patients with documented Gilbert's syndrome (unconjugated hyperbilirubinemia) bilirubin must be < 3 x ULN for age (patients with solid tumors)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN. (if liver metastases present =< 5 x ULN). For the purpose of this study, the ULN for ALT is 45 U/L regardless of baseline and the ULN for AST is 50 U/L regardless of baseline (patients with solid tumors)
* Serum albumin >= 2.5 g/dL (patients with solid tumors)
* International normalized ratio (INR)/prothrombin time (PT) and either partial thromboplastin or activated partial thromboplastin time (aPTT) =< 1.5 x ULN (patients with solid tumors)
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by either an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before Step 1 enrollment
* Corrected QT interval (QTc) prolongation to < 470 ms (females) or < 450 ms (males) based on average triplicate 12-lead electrocardiogram (ECG)
* Pulse oximetry > 93% on room air
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled as evidenced by no increase in seizure frequency in the prior 7 days
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v]5) resulting from prior chemotherapy, surgery, and/or radiation must be =< grade 2, with the exception of decreased tendon reflex (DTR). Any grade of DTR is eligible
* All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Pregnant, planning to become pregnant, or breast-feeding women will not be entered on this study because there is yet no available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method (e.g., male or female condom) for the duration of the study and upon completion of the study and for at least 7 months for females and 4 months for males after the last dose of study drug. Abstinence is an acceptable method of birth control

  * Methods considered as highly effective methods of contraception include:

    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

      * Oral
      * Intravaginal
      * Transdermal
    * Progestogen-only hormonal contraception associated with inhibition of ovulation:

      * Oral
      * Injectable
      * Implantable
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomized partner
    * Complete sexual abstinence defined as refraining from heterosexual intercourse. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception
* Non-child-bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle-stimulating hormone [FSH] > 40 mIU/mL and estradiol < 40 pg/mL [< 147 pmol/L] is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Male subjects must not freeze or donate sperm starting at Screening and throughout the study period, and at least 4 months after the final study drug administration. Preservation of sperm should be considered prior to enrolment in this study
* Female subjects must not donate, or retrieve for their own use, ova from the time of Screening and throughout the study treatment period, and for at least 7 months after the final study drug administration
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients who are receiving chloroquine or hydroxychloroquine within 14 days are not eligible for this trial
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with a medical history of myocardial infarction within 180 days before enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV) or troponin levels consistent with myocardial infarction as defined according to the manufacturer 28 days prior to enrollment are not eligible
* Patients who have a pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART) are not eligible
* Patients who have spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms are not eligible
* Patients with a known history of severe hypersensitivity to DS-8201a or any excipient contained in the DS-8201a drug formulation are not eligible
* Patients who have an uncontrolled infection or non-healing surgical site are not eligible
* Patients with a known history of substance abuse or any other clinically significant medical conditions (i.e. psychological conditions) that may, in the opinion of the investigator, interfere with the patient's participation in the clinical study or evaluation of the clinical study results are not eligible
* Patients who have pulmonary compromise, ex hypoxia, resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e. pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion etc.), or prior pneumonectomy are not eligible
* Patients who have a history of (non-infectious) ILD (interstitial lung disease)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening are not eligible
* Patients who have a pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or cell-free and concentrated ascites reinfusion therapy (CART) are not eligible. (Drainage and CART are not allowed within 2 weeks prior to screening assessment)
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival of DS-8201A for HER2+ osteosarcoma | At 24 weeks
  Frequency (%) of evaluable patients who are event-free after 24 weeks (4-months) of therapy.

SECONDARY OUTCOMES:
Incidence of adverse events of DS-8201A for HER2+ osteosarcoma | Up to 6 months
  Frequency (%) of evaluable patients with >= Grade 3 toxicity that is at least possibly related to the study agent stratified by dose level, part, and cycle (Cycle 1 vs. > Cycle 1).
Time to progression of DS-8201A for HER2+ osteosarcoma | Up to 1 year
  Median (95% CI) time-to-progression estimated by Kaplan-Meier curves by dose level.
Overall survival of DS-8201A for HER2+ osteosarcoma | Up to 1 year
  Median (95% CI) time-to-death estimated by Kaplan-Meier curves by dose level.
Event free survival of DS-8201A for HER2+ osteosarcoma | Up to 1 year
  Median (95% CI) time-to-event estimated by Kaplan-Meier curves by dose level.
Response rates of DS-8201A for HER2+ osteosarcoma | Up to 1 year
  The percent of responders will be estimated with 95% confidence intervals. Will be calculated as the percent of evaluable patients who are responders, and confidence intervals will be constructed accounting for the two-stage design.
Duration of response | Up to 1 year
  The duration of overall response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Damon R Reed, Principal Investigator — Pediatric Early Phase Clinical Trial Network
Locations (28):
- United States (28):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm